CLINICAL TRIAL: NCT06990841
Title: A Prospective Comparison of Two Different Sperm Preparation Techniques on the Prescence of DNA Fragmentation and Embryo Development
Brief Title: Comparison of Two Different Sperm Processing Methods and Their Effects on Sperm DNA Fragmentation and Embryo Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Kordus, PhD, HCLD (ABB) (Other)
Responsible Party: Sponsor-Investigator, Richard Kordus, PhD, HCLD (ABB), Director of ART Laboratories, Prisma Health-Upstate
Organization: Prisma Health-Upstate (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2295231-1
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: DNA Damage; DNA Strand Breaks; Sperm DNA Fragmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Gradient/swim-up vs Lenshooke CA0 device comparison (Experimental)
  Interventions: Device: sperm separation device

INTERVENTIONS:
Device: sperm separation device — comparison of DNA damage between the 2 interventions and subsequent embryo development and pregnancy rates

SUMMARY:
The goal of this clinical trial is to learn if the LensHooke CA0 device lowers DNA fragmentation in sperm samples compared to a gradient/swim-up technique.

The main questions it aims to answer are:

1. Does the LensHooke® CA0 device reduce DNA fragmentation compared to the gradient/swim-up technique?
2. Does the LensHooke® CA0 device improve concentration, motility, and morphology compared to the gradient/swim-up technique?
3. Is sibling embryo fertilization and development the same?
4. Are pregnancy rates different between the 2 groups?

1 semen sample will be split between the 2 treatment techniques. Half of the partner's egg cohort will be injected via intra-cytoplasmic sperm using sperm processed by one technique and the other half of the cohort will be injected by the sperm processed by the other technique. Both methods will look at DNA fragmentation, concentration, motility, and morphology of the sperm. Both methods will be compared in the resulting embryos looking at fertilization, embryo development and pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Samples with ≥15 M/mL spermatozoa concentration
* Female partner between 18 and 34 years old.
* Minimum of 4 fertilized eggs in gradient/swim prep group and 4 fertilized eggs in the Lenshooke prep group for each patient

Exclusion Criteria:

* Samples with <15 M/mL spermatozoa concentration
* female partner >35 years old
* female patient with recurrent pregnancy loss
* female patient with diminished ovarian reserve

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of sperm with DNA fragmentation | From enrollment until day after sample collection, approximately 1 month
  The method is based on the Sperm Chromatin Dispersion (SCD) test (Fernández et al., J. Androl 24:59-66, 2003; Fertil Steril 84:833-842, 2005). Intact unfixed spermatozoa (fresh, frozen/unthawed, diluted or neat samples) are immersed in an inert agarose microgel on a pretreated slide. An initial acid treatment denatures DNA in those sperm cells with fragmented DNA. Following this, the lysing solution removes most of the nuclear proteins, and in the absence of massive DNA breakage produces nucleoids with large halos of spreading DNA loops, emerging from a central core. However, the nucleoids from spermatozoa with fragmented DNA either do not show a dispersion halo or the halo is minimal. Slides are stained with Wright's stain. A minimum of 300 sperm per sample will be counted. The percentage of sperm with fragmented DNA will be calculated by dividing the sperm with small and no halos (fragmented sperm) by the total number of sperm counted.

SECONDARY OUTCOMES:
Concentration of sperm per mL | From enrollment until day after sample collection, approximately 1 month
  Assessed using a sperm class analyzer - SCA (CASA system) for sperm count. Semen samples will be loaded into 20 microliter depth fixed volume slides. Slides will be placed on the Microoptics SCA machine. Videos will be captured of fields until at least 200 motile sperm are captured. Concentration will be analyzed by counting the number of sperm within each field, corrected for the depth of the chamber, and multipled by the volume of the sample. Concentrations between fields will not vary by more than 15%.

OTHER OUTCOMES:
Percentage of motile sperm | From enrollment until day after sample collection, approximately 1 month
  Assessed using a sperm class analyzer - SCA (CASA system) for sperm motility. Semen samples will be loaded into 20 microliter depth fixed volume slides. Slides will be placed on the Microoptics SCA machine. Videos will be captured of fields until at least 200 motile sperm are captured. Motility will be calculated as the number of motile sperm counted divided by the total number of sperm counted. Types of motility will be noted according to WHO semen analysis groupings, hyperactivation, and kinetic motion parameters.
Percentage of Sperm with normal morphology Using Kruger Strict Criteria | From enrollment until day after sample collection, approximately 1 month
  10 uL volumes of sperm samples will be placed on pre-stained morphology slides using methylene blue/cresyl violet stain. A minimum of 200 sperm will be counted and assessed for normal vs abnormal sperm morphology using Kruger strict criteria. Percentage of normal sperm will be assessed my dividing the number of normal sperm by the total number of sperm counted.
Percentage of egg fertilization | From enrollment until a week after sample collection, approximately 5 weeks
  The number of fertilized eggs (zygotes) will be divided by the number of eggs inseminated
Numerical score of morphokinetic embryo development | From enrollment until a week after sample collection, approximately 5 weeks
  Embryo development will be monitored using a time-lapse incubator. A score will be generated based on when the embryos meets developmental time points. The embryo will receive 2 points for each time point it successfully completes with expected parameters. Embryos will receive 1 point for each time point it completes but outside the expected time parameters. i.e. if an embryo has the first cleavage between 23-25 hours it will receive 2 points. If it cleaves earlier than 23 hours or later than 25 hours it will receive 1 point. The total score an embryo receives will be tallied from the time of insemination until the embryo is frozen.
Qualitative embryo grade | From enrollment until a week after sample collection, approximately 5 weeks
  All embryos will be graded according to a 3-part grading scale at the time of cryopreservation between days 5 and 7 of culture. The embryo will be given a number score of 1-6 based on the embryo's size, size of the blastocoel fluid cavity, and whether or not it is inside, hatching out, or completely hatched out the zona. Each embryo will get a letter grade for the quality of the inner cell mass either A, B, C, or D. Each embryo will get a second letter grade for the quality of the trophectoderm A, B, C, or D.
Percentage of patients that become pregnant and deliver a baby | From enrollment until a delivery of infant, up to 18 months
  Calculated by the number of patients that become pregnant (assessed by the presence of a fetal heartbeat 5-6 weeks following embryo transfer) divided by the total number of embryos transferred. Live birth will be calculated by the number of patients that give birth divided by the number of embryos transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kordus, PhD, Principal Investigator — Prisma Health-Upstate Fertility Center of the Carolinas
Locations (1):
- Prisma Health-Upstate Fertility Center of the Caroliinas, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho CLT, Vaughan-Constable DR, Ramsay J, Jayasena C, Tharakan T, Yap T, Whiteman I, Graham N, Minhas S, Homa ST. The relationship between genitourinary microorganisms and oxidative stress, sperm DNA fragmentation and semen parameters in infertile men. Andrologia. 2022 Mar;54(2):e14322. doi: 10.1111/and.14322. Epub 2021 Nov 24. PMID 34817086
- [Background] Amor H, Hammadeh ME, Mohd I, Jankowski PM. Impact of heavy alcohol consumption and cigarette smoking on sperm DNA integrity. Andrologia. 2022 Aug;54(7):e14434. doi: 10.1111/and.14434. Epub 2022 Apr 28. PMID 35484935
- [Background] Cho CL, Agarwal A, Majzoub A, Esteves SC. Clinical utility of sperm DNA fragmentation testing: concise practice recommendations. Transl Androl Urol. 2017 Sep;6(Suppl 4):S366-S373. doi: 10.21037/tau.2017.07.28. PMID 29082146
- [Background] Rex AS, Aagaard J, Fedder J. DNA fragmentation in spermatozoa: a historical review. Andrology. 2017 Jul;5(4):622-630. doi: 10.1111/andr.12381. PMID 28718529